CLINICAL TRIAL: NCT00477126
Title: Bioequivalence Study of Generic GPO Ritonavir Versus Norvir® in Thai Healthy Volunteers
Brief Title: Bioequivalence Study of Generic GPO Ritonavir Versus Norvir®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: The Government Pharmaceutical Organization (Other Government)
Responsible Party: Kiat Ruxrungtham, HIV-NAT
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HIV-NAT 037
Record Dates: First submitted 2007-05-20; First posted 2007-05-22 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: ritonavir generic capsule; Norvir®; Thailand; Determine bioequivalence between Norvir and GPO ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): start generic product cross over to reference product
  Interventions: Drug: GPO ritonavir versus Norvir
- 2 (Active Comparator): start reference product cross over to generic product
  Interventions: Drug: GPO ritonavir versus Norvir

INTERVENTIONS:
Drug: GPO ritonavir versus Norvir — RTV generic compared to reference drugs (Norvir, Abbott)

SUMMARY:
To establish bioequivalence of ritonavir generic capsule, with Norvir® as reference drug.

DETAILED DESCRIPTION:
This study will be performed to evaluate if the new generic GPO ritonavir product is bio-equivalent to Norvir and to compare the short-term tolerability and safety profiles.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Healthy male or female 18-45 years old
* Documented negative test for HIV-1 infection < 1 wk prior to start of study and with no risk of
* HIV exposure in the last 6 months
* For female subjects: documented negative pregnancy test <3 wk prior to start of study, not breastfeeding
* BMI 18-25
* Normal physical examination
* Normal CBC, BUN, Cr, AST, ALT, Total bilirubin, no evidence of active or chronic HBV or HCV Infection

Exclusion Criteria:

* History of sensitivity/idiosyncrasy to the drug or chemically related compounds or excipients, which may be employed in the study.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* Inability to understand the nature and extent of the study and the procedures required.
* Participation in a drug study within 60 days prior to the first dose.
* Febrile illness within 3 days before the first dose.
* Use of concomitant medication
* Smoke cigarettes not more than 10 cigarettes a day.
* Drink alcohol not more than 2 units a day
* Discontinue smoking and alcohol for at least 1 month before enrollment.
* Take other medication regularly
* Involvement in any drug addiction
* Heart disease, hypertension, liver disease, kidney disease, GI disease, allergic disease or other diseases which may interfere with the PK of study drugs

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2007-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Establish bioequivalence of generic GPO ritonavir, with Norvir® as the reference drug. | 2 months

SECONDARY OUTCOMES:
Evaluate the short-term tolerability and safety profiles of generic ritonavir in healthy male and female volunteers. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT)
Locations (1):
- The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT), Bangkok, Bangkok, Thailand

REFERENCES:
- See also: The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org